CLINICAL TRIAL: NCT06398821
Title: A Dose Ranging Target Engagement Study of a Food-Grade Pectic Food Supplement (G3P-01) in Volunteers With Elevated Levels of Galectin-3 - the Galaxy Study
Brief Title: G3P-01 in Volunteers With Elevated Galectin-3
Acronym: Galaxy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: General Practitioners Research Institute (Network)
Collaborators: G3 Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: GPRI-23001-G3P
Record Dates: First submitted 2023-08-23; First posted 2024-05-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-04

CONDITIONS: Galectin 3; Healthy Aging
Keywords: Galectin 3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo for 30 days
  Interventions: Dietary Supplement: Placebo
- G3P-01 100mg (Active Comparator): G3P-01 100mg daily for 30 days
  Interventions: Dietary Supplement: G3P-01
- G3P-01 250mg (Active Comparator): G3P-01 250mg daily for 30 days
  Interventions: Dietary Supplement: G3P-01
- G3P-01 1000mg (Active Comparator): G3P-01 1000mg daily for 30 days
  Interventions: Dietary Supplement: G3P-01

INTERVENTIONS:
Dietary Supplement: G3P-01 — Nutritional supplement to promote healthy aging
  Arms: G3P-01 1000mg; G3P-01 100mg; G3P-01 250mg
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
G3P-01 is an investigational pectin extracted, enriched and purified from commercial squash puree intended for human consumption. Pectins are an important constituent of fruits and vegetables, and health benefits are attributed to its intake. Some of the health benefits of pectins are attributed to inhibition of galectin-3. This study investigates if 30-days of G3P-01 intake in individuals with elevated galectin-3 induces biomarker changes that can be attributed to target engagement. Participants will be randomized into four groups (placebo, 100mg, 250mg and 1000mg G3P-01).

ELIGIBILITY:
Inclusion Criteria:

* Invited through cohort study.
* Plasma galectin-3 level of 16 ng/mL or higher
* Male and female subjects ≥45 and ≤75 years of age
* Females will be non-pregnant, non-lactating, and have no intent to become pregnant during the study period.
* Able to participate in the study in the opinion of the Investigator.
* Has the ability to understand the requirements of the study and is willing to comply with all study procedures.
* An Independent Ethics Committee or in Dutch Medisch- Ethische Toetsingscommissie (METC) -approved informed consent is signed and dated prior to any study-related activities.

Exclusion Criteria:

* Existing clinically significant concurrent medical condition which in the opinion of the Investigator may interfere with the study.
* Clinically significant abnormal laboratory test values, as determined by the Investigator, at Screening.
* Participation in a clinical trial of an investigational drug within 30 days prior to Screening, or is currently participating in another trial of an investigational drug, supplement or device.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
To evaluate target engagement attributable to G3P-01 use in volunteers with elevated galectin-3 (≥ 16.0ng/mL) | 4 months
  Change from baseline of pathway markers consistent with galectin-3 inhibition (dose-response effect) measured by proteomics
To evaluate tolerability of G3P-01 | 4 months
  Changes in the Gastrointestinal Symptom Rating Scale (1 means no symptoms, 7 means symptoms)
To evaluate tolerability of G3P-01 | 4 months
  Number of participants with abnormal laboratory tests results
To evaluate tolerability of G3P-01 | 4 months
  Number of participants with abnormal physical examination findings

CONTACTS AND LOCATIONS:
Overall Officials: J WH Kocks, MD, PhD, Principal Investigator — General Practitioners Research Institute
Locations (1):
- General Practitioners Research Institute, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No